CLINICAL TRIAL: NCT05769530
Title: Dexmedetomidine Combined With Nalbuphine Advanced Analgesia on the Quality of Recovery After General Anesthesia in Elderly Patients
Brief Title: Advanced Analgesia on the Quality of Recovery After General Anesthesia in Elderly Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lili Jia (Other)
Responsible Party: Sponsor-Investigator, Lili Jia, sponsor, Tianjin First Central Hospital
Organization: Tianjin First Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023TJY
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: General Anesthetics，Emergence Agitation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- DEX and Nalbuphine group (Experimental): In group B, DEX 0.5μg/kg was injected intravenously 30min before the end of the operation, 30min after the pump, and Nalbuphine 0.20 mg/kg (5 mL) was injected intravenously 30min before the end of the operation.
  Interventions: Drug: Nalbuphine，dexmedetomidine
- placebo group (Placebo Comparator): Group A was continuously injected with normal saline during the operation, and 5 mL of normal saline was injected intravenously 30min before the end of the operation
  Interventions: Drug: Nalbuphine，dexmedetomidine
- nalbuphine group (Experimental): Group C was continuously injected with normal saline 30 minutes before the end of the operation, and intravenous injection of nalbuphine 0.20 mg/kg (5 mL) 30 minutes before the end of the operation.
  Interventions: Drug: Nalbuphine，dexmedetomidine

INTERVENTIONS:
Drug: Nalbuphine，dexmedetomidine — According to the drug use, the subjects were divided into group A, which was continuously injected with normal saline during the operation, and intravenously injected with 5 mL normal saline 30 minutes before the end of the operation. In group B, DEX 0.5μg/kg was injected intravenously during the operation, which was completed in 10 min, and Nalbuphine 0.20 mg/kg (5 mL) was injected intravenously 30min before the end of the operation. After the operation, all anesthetic drugs were stopped and the patient was transferred to PACU with intubation.

SUMMARY:
Recovery period of general anesthesia refers to the period from the end of anesthesia infusion to recovery of the patient after the operation. In patients with general anesthesia, the depth of anesthesia is reduced in the early stage of recovery, the cerebral cortex is still in a state of inhibition, and the subcortical center is often in a state of high sensitivity to external stimulation. At this time, due to drug effects, pain, hypoxemia, undetected aspiration, pneumothorax, urinary retention, tracheal catheter stimulation, urinary tube stimulation and other factors, the patient will be induced to appear restless reaction, and cause drastic changes in hemodynamics. Especially for the elderly with organ dysfunction, it may increase postoperative complications, prolong hospital stay and increase hospital costs.

DETAILED DESCRIPTION:
In recent years, a number of studies have shown that dexmetropil and nalbuphine can reduce postoperative agitation and cough during extubation, respectively, without increasing extubation time. Nalbuphine is a combination of opioid receptor excitation-antagonistic analgesic, which can be combined with μ, κand δ receptors. Nalbuphine has complete excitatory effect on κreceptor and partial antagonistic effect on μ receptor, so it has analgesic and sedative effect. Its analgesic intensity is similar to that of morphine, which can be used to relieve moderate to severe pain and also reduce visceral pain. With little addiction, it can effectively prevent anesthetic stimulation caused by surgical trauma and reduce intraoperative inflammation. Nalbuphine has few cardiovascular side effects, mild respiratory depression and capping effect. As with other agonist antagonists, nabulphine interferes with the adverse reactions associated with pure μ-receptor agonists, such as nausea, vomiting, and pruritus. Dexmedetomidine belongs to an agonist of α2 adrenergic receptor, which has analgesic, sedative, antianxiety, stable kinetics and reducing stress response. It can activate the α2 receptor in the patient's body, thus inhibiting the release of norepinephrine in the patient's body, and then play a role in analgesia, sedation, anti-anxiety.

The main result of this study was the occurrence of agitation within 30 minutes after general anesthesia. The occurrence of agitation was determined by the Riker sedation-excitement score (5-7).

Secondary research indicators:

1. EA occurred 0, 10, 20, 30 minutes after extubation by PACU.
2. Chills occurred 0, 10, 20, 30 minutes after extubation in PACU.
3. Postoperative pain was assessed by visual analogue scale (VAS) at 0, 10, 20 and 30min after extubation by PACU.
4. Classification of choking degree within 30 minutes after extubation after recovery
5. The changes of vital signs (heart rate, blood pressure and oxygen saturation) were observed at 0min, 10min, 20min and 30min after extubation.
6. extubation time: the time from anesthetic withdrawal to extubation.
7. Length of hospital stay in PACU: the duration from the end of the operation to the exit of PACU.
8. Oxygenation index: The radial artery blood was taken for blood gas analysis before incision, after surgery and 5 minutes after extubation, and the oxygenation index (PaO2/FiO2) was calculated.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥60, gender unlimited;

  (2) ventilator assisted ventilation after endotracheal intubation;

  (3) General anesthesia surgery;

Exclusion Criteria:

* (1) Allergy to the drugs used in this study;

  (2) any sedative, analgesic, antiemetic or antipruritic drugs taken 24 hours before the operation;

  (3) History of severe bradycardia (heart rate < 50 beats/min);

  (4) moderate to severe hepatic and renal dysfunction;

  (5) Patients with neurological diseases;

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
The main outcome of this study was the occurrence of agitation from the time of awakening to 30 minutes after extubation | from the time of awakening to 30 minutes after extubation
  Riker sedation-excitement score, 5 to 7 points to determine the occurrence of agitation.

SECONDARY OUTCOMES:
postoperation pain | from the time of awakening to 30 minutes after extubation
  Postoperative pain was assessed by visual analogue scale (VAS) at 0, 10, 20 and 30min after extubation by PACU.
Postoperative cough | from the time of awakening to 30 minutes after extubation
  Grade of choking

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - TianJin First Central Hospital, Tianjin, Tianjin Municipality
  - Tian Jin First Center Hospital, Tianjin

DOCUMENTS (1):
  • Study Protocol (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT05769530/Prot_000.pdf